CLINICAL TRIAL: NCT05628103
Title: An 8-Week, Open-Label Study Evaluating the Effectiveness, Safety and Tolerability of SEP-363856 in Subjects With Schizophrenia Switched From Typical or Atypical Antipsychotic Agents
Brief Title: A Clinical Study That Will Evaluate How Well SEP-363856 Works and How Safe it is in People With Schizophrenia That Switch to SEP-363856 From Their Current Antipsychotic Medication
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Otsuka Pharmaceutical Development & Commercialization, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: SEP361-308
Record Dates: First submitted 2022-11-16; First posted 2022-11-28 (Actual); Results first posted 2025-11-12 (Actual); Last update posted 2025-12-11 (Actual); Status verified 2025-03

CONDITIONS: Schizophrenia
Keywords: Schizophrenia
MeSH Terms: conditions — Schizophrenia | interventions — SEP-363856

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- SEP-363856 (Experimental): Participants received flexible doses of SEP-363856 50 to 100 milligrams per day (mg/day), orally, once daily (QD) up to Week 8. The dose was titrated up from 50 mg/day on Days 1 to 3, to 75 mg/day on Days 4 to 7. Beginning Day 8, the dose was adjusted within the range of 50 mg/day to 100 mg/day in 25 mg increments (i.e. 50, 75, or 100 mg/day) up to Week 8.
  Interventions: Drug: SEP-363856

INTERVENTIONS:
Drug: SEP-363856 — SEP-363856 flexibly dosed for 8 weeks.

SUMMARY:
This study evaluated how well SEP-363856 works and how safe it is in people with schizophrenia that switch to SEP-363856 from their current antipsychotic medication.

DETAILED DESCRIPTION:
This was an 8-week, outpatient, multicenter, open-label, single-group, flexible-dose study.

Following a screening period of up to 21 days, eligible participants took part in the study. In the 8-week treatment period, participants were treated with SEP-363856 while continuing to take the full dose of their pre-switch antipsychotic. After the end of the treatment period, participants were required to complete the follow-up visit, 7 days after the last dose of SEP-363856.

ELIGIBILITY:
Inclusion Criteria: This list is not all inclusive

* Participants meets Diagnostic and Statistical Manual of Mental Disorders, Fifth Edition (DSM-5) criteria for a diagnosis of schizophrenia.
* Participants are judged to be clinically stable (ie, no evidence of an acute exacerbation of schizophrenia) by the Investigator for at least 8 weeks prior to Baseline.
* Participants must be judged by the Investigator to be an appropriate candidate for switching current antipsychotic medication due to safety or tolerability concerns and/or insufficient efficacy.
* Participants are taking an oral antipsychotic and the antipsychotic regimen has been stable for at least 6 weeks prior to Screening.

Exclusion Criteria:This list is not all inclusive

* Participant has a current DSM-5 diagnosis or presence of symptoms consistent with a major psychiatric disorder, other than schizophrenia, that is the primary focus of treatment.
* Participants are at significant risk of harming self or others based on investigator's judgment.
* Participant has any clinically significant unstable medical condition or any clinically significant chronic disease that in the opinion of the Investigator, would limit the participant's ability to complete and/or participate in the study.
* Female participant who is pregnant or lactating.
* Participant tests positive for drugs of abuse at Screening.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 101 (Actual)
Dates: Start 2022-12-19 (Actual); Primary Completion 2024-04-01 (Actual); Study Completion 2024-04-01 (Actual)

CONTACTS AND LOCATIONS:
Locations (25):
- United States (25):
  - Advanced Research Center, Inc., Anaheim, California
  - Clinical Innovations Inc., Bellflower, California
  - ProScience Research Group, Culver City, California
  - Collaborative Neuroscience Research, LLC, Garden Grove, California
  - Synergy San Diego, Lemon Grove, California
  - Clinical Innovations, Inc, Riverside, California
  - California Neuropsychopharmacology Clinical Research Institute, LLC (CNRI-San Diego, LLC), San Diego, California
  - CMB Clinical Trials, Santee, California
  - Cenexel CNS Research, Torrance, California
  - Larkin Behavioral Health Services, Hollywood, Florida
  - Premier Clinical Research Institute, Inc., Miami, Florida
  - Wellness Research Center, Miami, Florida
  - Nova Psychiatry, Inc., Orlando, Florida
  - Advanced Discovery Research LLC, Atlanta, Georgia
  - Atlanta Center for Medical Research, Atlanta, Georgia
  - Atlanta Behavioral Research, Atlanta, Georgia
  - Uptown Research, Chicago, Illinois
  - CBH Health, Gaithersburg, Maryland
  - PsychCare Consultants Research, St Louis, Missouri
  - IMA Clinical Research, Las Vegas, Nevada
  - Hassman Research Institute, Berlin, New Jersey
  - New Hope Clinical Research, Charlotte, North Carolina
  - Clinical Trials of America, LLC, Hickory, North Carolina
  - Charak Clinical Research Center, Garfield Heights, Ohio
  - Pillar Clinical Research, LLC, Richardson, Texas

IPD SHARING:
Plan to Share IPD: Yes
Anonymized Individual participant data (IPD) that underlie the results of this study will be shared with researchers to achieve aims pre-specified in a methodologically sound research proposal. Small studies with less than 25 participants are excluded from data sharing.
Supporting Information: Study Protocol, SAP, ICF
Time Frame: Data will be available after marketing approval in global markets, or beginning 1-3 years following article publication. There is no end date to the availability of the data.
Access Criteria: Otsuka will share data on the Vivli data sharing platform which can be found here: https://vivli.org/ourmember/Otsuka/
URL: http://clinical-trials.otsuka.com

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants took part in the study at 26 clinical sites in the United States (US) from 19 December 2022 to 01 April 2024.
Pre-assignment Details: A total of 243 participants were screened, of which 101 participants entered the study, and all 101 participants received at least one dose of SEP-363856 in the 8-week treatment period.
Period: Overall Study
Arm/Group | SEP-363856
Started | 101
Safety Population | 101
Completed | 83
Not Completed | 18
Not completed — Adverse Event | 7
Not completed — Withdrawal by Subject | 3
Not completed — Lost to Follow-up | 3
Not completed — Lack of Efficacy | 1
Not completed — Non-Compliance With Study Drug | 4

BASELINE CHARACTERISTICS:
Population: Safety population included all participants that were enrolled and received the study drug.
Groups:
- SEP-363856: Participants received flexible doses of SEP-363856 50 to 100 mg/day, orally, QD up to Week 8. The dose was titrated up from 50 mg/day on Days 1 to 3, to 75 mg/day on Days 4 to 7. Beginning Day 8, the dose was adjusted within the range of 50 mg/day to 100 mg/day in 25 mg increments (i.e. 50, 75, or 100 mg/day) up to Week 8.
Arm/Group | SEP-363856
Number analyzed (Participants) | 101
Age, Continuous [Mean (Standard Deviation); unit: years] | 48.1 (12.02)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 29
  Male | 72
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 18
  Not Hispanic or Latino | 83
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 3
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 64
  White | 32
  More than one race | 1
  Unknown or Not Reported | 1

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants Who Discontinued From the Study Due to Clinical Reasons
Description: Discontinuation for clinical reasons was defined as reasons due to adverse event (AE) or lack of efficacy. AEs are defined as untoward medical occurrences that started at the same time of or after the first dose of study drug. The percentage of participants who discontinued for clinical reasons was calculated by a proportion consisting of the number of participants who experience a discontinuation event due to clinical reasons as the numerator divided by the number of participants in the safety population as the denominator multiplied by 100 along with a corresponding 95% confidence interval (CI). 95% CI was calculated using the normal approximation method.
Time Frame: From the first dose of the study drug up to end of follow up (up to Week 9)
Population: Safety population included all participants that were enrolled and received the study drug. Percentages are rounded off to the nearest decimal point.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | SEP-363856
Number analyzed (Participants) | 101
percentage of participants | 7.9 [2.7 to 13.2]

2. Secondary Outcome: Percentage of Participants Who Discontinued From the Study Due to Any Reason
Description: The percentage of participants who discontinued from the study due to any reason was calculated by a proportion consisting of the number of participants who experience a discontinuation event due to any reason as the numerator divided by the number of participants in the safety population as the denominator multiplied by 100 along with a corresponding 95% CI. 95% CI was calculated using the normal approximation method.
Time Frame: From first dose of the study drug up to end of follow-up period (up to Week 9)
Population: as for outcome 1
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | SEP-363856
Number analyzed (Participants) | 101
percentage of participants | 17.8 [10.4 to 25.3]

ADVERSE EVENTS:
Time Frame: From first dose of study drug up to end of follow up period (up to Week 9)
Description: Safety population included all participants that were enrolled and received the study drug.
Arm/Group | SEP-363856
All-Cause Mortality (participants affected / at risk) | 0/101
Serious Adverse Events (participants affected / at risk) | 4/101
Other Adverse Events (participants affected / at risk) | 13/101
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | SEP-363856 (N=101)
Schizophrenia (Psychiatric disorders) | 4
OTHER ADVERSE EVENTS (reported when occurring in more than 2% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | SEP-363856 (N=101)
Dry mouth (Gastrointestinal disorders) | 3
Nausea (Gastrointestinal disorders) | 3
Dizziness (Nervous system disorders) | 5
Insomnia (Psychiatric disorders) | 4

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol (2023-11-06): https://cdn.clinicaltrials.gov/large-docs/03/NCT05628103/Prot_000.pdf
  • Statistical Analysis Plan (2024-05-06): https://cdn.clinicaltrials.gov/large-docs/03/NCT05628103/SAP_001.pdf